CLINICAL TRIAL: NCT04532606
Title: Impact of Remimazolam Tosilate for General Anesthesia on Prognosis After Bladder Cancer Surgery: a Randomized Controlled Trial
Brief Title: Impact of Remimazolam on Prognosis After Bladder Cancer Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other); Navy General Hospital, Beijing (Other); Guizhou Provincial People's Hospital (Other); Jiangsu Provincial People's Hospital (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-212
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Benzodiazepines; Bladder Cancer; Delirium; Surgery; Cancer Recurrence
Keywords: Remimazolam; Bladder Cancer; Surgery; Emergence Delirium; Recurrence-free Survival
MeSH Terms: conditions — Urinary Bladder Neoplasms; Delirium; Emergence Delirium | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Remimazolam is administered intravenously for anesthesia induction and maintenance. The dose and infusion rate is adjusted to maintain Bispectral Index (BIS) value between 40 and 60. Analgesia is maintained with remifentanil and/or sufentanil. Muscle relaxation is maintained with rocuronium and/or cisatracurium. Sevoflurane inhalation is provided when considered necessary.
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): Propofol is administered intravenously for anesthesia induction and maintenance. The dose and infusion rate is adjusted to maintain BIS value between 40 and 60. Analgesia is maintained with remifentanil and/or sufentanil. Muscle relaxation is maintained with rocuronium and/or cisatracurium. Sevoflurane inhalation is provided when considered necessary.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is administered intravenously for anesthesia induction and maintenance. The dose and infusion rate is adjusted to maintain BIS value between 40 and 60. Analgesia is maintained with remifentanil and/or sufentanil. Muscle relaxation is maintained with rocuronium and/or cisatracurium. Sevoflurane inhalation is provided when considered necessary.
  Other Names: Remimazolam anesthesia
  Arms: Remimazolam group
Drug: Propofol — Propofol is administered intravenously for anesthesia induction and maintenance. The dose and infusion rate is adjusted to maintain BIS value between 40 and 60. Analgesia is maintained with remifentanil and/or sufentanil. Muscle relaxation is maintained with rocuronium and/or cisatracurium. Sevoflurane is provided when considered necessary.
  Other Names: Propofol anesthesia
  Arms: Propofol group

SUMMARY:
Bladder cancer is one of the most common genitourinary cancers. Transurethral resection of bladder tumor (TURBT) is the standard therapy for nonmuscle invasive bladder cancer. However, patients after TURBT are at risk for recurrence and progression. Benzodiazepines are proved to inhibit proliferation of multiple types of cancer cells in vitro. Delirium is an acute onset and transient cerebral dysfunction and is associated with worse outcomes. Previous studies indicated that benzodiazepines increase incidence of postoperative delirium. Remimazolam is a new benzodiazepine with rapid onset and ultra-short activity. The aims of this study are to explore the impact of remimazolam for general anesthesia on emergency delirium and recurrence-free survival in patients undergoing bladder cancer surgery.

DETAILED DESCRIPTION:
Bladder cancer is one of the most common genitourinary cancers. Approximately 70-80% of bladder cancers are nonmuscle invasive, including those of Ta-T1 stage and carcinoma in situ. Transurethral resection of bladder tumor (TURBT) is the standard therapy for nonmuscle invasive bladder cancer. However, patients after TURBT are at a high risk of recurrence and progression.

Recently, impacts of anesthetic agents on tumor cells have attracted more attention. Benzodiazepines are found to inhibit proliferation of lymphoma, neural tumor, lung cancer, rectal cancer and breast cancer cells in vitro. Midazolam may have anti-tumor effects through induction of apoptosis and inhibition of inflammatory reaction. However, clinical evidence regarding effects of benzodiazepines on outcomes after cancer surgery remains lacking.

Remimazolam is a new benzodiazepine with rapid onset and ultra-short activity. It is rapidly metabolized by tissue esterases to inactive metabolite and can be reversed by flumazenil. Therefore, patients wake up rapidly even after prolonged infusions. It is also found to produce less respiratory and circulatory depression when compared with propofol.

Delirium is an acute onset and transient cerebral dysfunction, and is associated with worse outcomes including prolonged hospitalization, worse functional recovery, cognitive decline, and increased mortality rate. Previous studies indicated that benzodiazepines increase incidence of postoperative delirium, possibly due to prolonged action. With the property of ultra-short activity, remimazolam may not increase the incidence of delirium. But evidence is lacking in this aspect.

The aims of this study are to explore the impact of remimazolam on emergency delirium and recurrence-free survival in patients undergoing bladder cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years and <90 years;
2. Preoperative diagnosis is non-muscle-invasive bladder cancer(Ta-T1);
3. Scheduled to undergo transurethral resection of bladder tumor;
4. Agree to participate, and provide written informed consent.

Exclusion Criteria:

1. Refuse to participate;
2. Emergent surgery;
3. Combined with other malignant tumors;
4. Use of benzodiazepines for 1 week within the last month before surgery;
5. Preoperative history of schizophrenia, epilepsy, parkinsonism or myasthenia gravis;
6. Inability to communicate in the preoperative period due to coma, profound dementia, language barrier, or end-stage disease;
7. Critical illness (preoperative American Society of Anesthesiologists physical status classification ≥IV), severe hepatic dysfunction (Child-Pugh class C), or severe renal dysfunction (undergoing dialysis before surgery);
8. The purpose of surgery is to make a diagnosis or preoperative judgement is that tumor cannot be completely removed.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence delirium (early). | Up to 2 hours during the stay in post-anesthesia care unit after surgery.
  Emergence delirium is assessed with the Confusion Assessment Method for the Intensive Care Unit at 10 and 30 minutes after admission to the post-anesthesia care unit after surgery.
Recurrence-free survival (long-term). | Up to 3 years after surgery.
  Time from surgery to recurrence/metastasis or all-cause death, whichever come first.

SECONDARY OUTCOMES:
Incidence of postoperative delirium (early). | During the first 3 days after surgery.
  Delirium is assessed twice daily with the Chinese version of the 3-minute diagnostic interview for Confusion Assessment Method-defined delirium.
Incidence of postoperative nausea and vomiting (early). | Up to 24 hours after surgery.
  Incidence of postoperative nausea and vomiting.
Incidence of intraoperative awareness (early). | Up to 1 day after surgery.
  Intraoperative awareness is assessed with modified Brice interview before discharge from the post-anesthesia care unit and on the 1st day after surgery. The interview included five questions: (1) What was the last thing you remembered happening before you went to sleep? (2) What is the first thing you remember after your operation? (3) Can you remember anything in between? (4) Can you remember if you had any dreams during your operation? (5) What was the worst thing about your operation?
Length of stay in hospital after surgery (early). | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of non-delirium complications (early). | Up to 30 days after surgery.
  Non-delirium complications are defined as newly occurred medical conditions other than delirium that are harmful for patients' recovery and required therapeutic intervention, i.e., grade 2 or higher on Clavien-Dindo classification.
All-cause 30-day mortality (early). | Up to 30 days after surgery.
  All-cause 30-day mortality.
Overall survival (long-term). | Up to 3 years after surgery.
  Time from surgery to all-cause death.
Event-free survival (long-term). | Up to 3 years after surgery.
  Time from surgery to serious events, cancer recurrence/metastasis, or all-cause death, whichever come first. Serious events are defined as any new onset disease that required hospitalization and/or surgical intervention.
Health related quality of life of 1-year survivors (long-term). | At the end of the 1st year after surgery.
  Health related quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

OTHER OUTCOMES:
Intensity of pain (early). | During the first 3 days after surgery.
  Assessed twice daily (8-10 am and 18-20 pm) with the Numeric Rating Scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain).
Subjective sleep quality (early). | During the first 3 days after surgery
  Assessed in the morning (8-10 am) with the Numeric Rating Scale (NRS; an 11-point scale where 0=the best sleep and 10=the worst sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Wang Dong-Xin, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (6):
- China (6):
  - Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality
  - The Sixth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijin, Bejing
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zheng R, Zhang S, Zeng H, Xia C, Zuo T, Yang Z, Zou X, He J. Cancer incidence and mortality in China, 2013. Cancer Lett. 2017 Aug 10;401:63-71. doi: 10.1016/j.canlet.2017.04.024. Epub 2017 May 3. PMID 28476483
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Soukup V, Capoun O, Cohen D, Hernandez V, Babjuk M, Burger M, Comperat E, Gontero P, Lam T, MacLennan S, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Sylvester R, Yuan Y, Zigeuner R. Prognostic Performance and Reproducibility of the 1973 and 2004/2016 World Health Organization Grading Classification Systems in Non-muscle-invasive Bladder Cancer: A European Association of Urology Non-muscle Invasive Bladder Cancer Guidelines Panel Systematic Review. Eur Urol. 2017 Nov;72(5):801-813. doi: 10.1016/j.eururo.2017.04.015. Epub 2017 Apr 28. PMID 28457661
- [Background] Allard P, Bernard P, Fradet Y, Tetu B. The early clinical course of primary Ta and T1 bladder cancer: a proposed prognostic index. Br J Urol. 1998 May;81(5):692-8. doi: 10.1046/j.1464-410x.1998.00628.x. PMID 9634043
- [Background] Holmgren L, O'Reilly MS, Folkman J. Dormancy of micrometastases: balanced proliferation and apoptosis in the presence of angiogenesis suppression. Nat Med. 1995 Feb;1(2):149-53. doi: 10.1038/nm0295-149. PMID 7585012
- [Background] Hofer SO, Molema G, Hermens RA, Wanebo HJ, Reichner JS, Hoekstra HJ. The effect of surgical wounding on tumour development. Eur J Surg Oncol. 1999 Jun;25(3):231-43. doi: 10.1053/ejso.1998.0634. PMID 10336800
- [Background] Eggermont AM, Steller EP, Marquet RL, Jeekel J, Sugarbaker PH. Local regional promotion of tumor growth after abdominal surgery is dominant over immunotherapy with interleukin-2 and lymphokine activated killer cells. Cancer Detect Prev. 1988;12(1-6):421-9. PMID 3263198
- [Background] Stevens MF, Werdehausen R, Gaza N, Hermanns H, Kremer D, Bauer I, Kury P, Hollmann MW, Braun S. Midazolam activates the intrinsic pathway of apoptosis independent of benzodiazepine and death receptor signaling. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):343-9. doi: 10.1097/AAP.0b013e318217a6c7. PMID 21701267
- [Background] Wang C, Datoo T, Zhao H, Wu L, Date A, Jiang C, Sanders RD, Wang G, Bevan C, Ma D. Midazolam and Dexmedetomidine Affect Neuroglioma and Lung Carcinoma Cell Biology In Vitro and In Vivo. Anesthesiology. 2018 Nov;129(5):1000-1014. doi: 10.1097/ALN.0000000000002401. PMID 30157038
- [Background] Mishra SK, Kang JH, Lee CW, Oh SH, Ryu JS, Bae YS, Kim HM. Midazolam induces cellular apoptosis in human cancer cells and inhibits tumor growth in xenograft mice. Mol Cells. 2013 Sep;36(3):219-26. doi: 10.1007/s10059-013-0050-9. Epub 2013 Sep 2. PMID 24008365
- [Background] Beinlich A, Strohmeier R, Kaufmann M, Kuhl H. Specific binding of benzodiazepines to human breast cancer cell lines. Life Sci. 1999;65(20):2099-108. doi: 10.1016/s0024-3205(99)00475-0. PMID 10579463
- [Background] Barends CRM, Absalom AR, Struys MMRF. Drug selection for ambulatory procedural sedation. Curr Opin Anaesthesiol. 2018 Dec;31(6):673-678. doi: 10.1097/ACO.0000000000000652. PMID 30124543
- [Background] Cornett EM, Novitch MB, Brunk AJ, Davidson KS, Menard BL, Urman RD, Kaye AD. New benzodiazepines for sedation. Best Pract Res Clin Anaesthesiol. 2018 Jun;32(2):149-164. doi: 10.1016/j.bpa.2018.06.007. Epub 2018 Jul 3. PMID 30322456
- [Background] Goudra BG, Singh PM. Remimazolam: The future of its sedative potential. Saudi J Anaesth. 2014 Jul;8(3):388-91. doi: 10.4103/1658-354X.136627. PMID 25191193
- [Background] Ilic RG. Fospropofol and remimazolam. Int Anesthesiol Clin. 2015 Spring;53(2):76-90. doi: 10.1097/AIA.0000000000000053. No abstract available. PMID 25807020
- [Background] Johnson KB. New horizons in sedative hypnotic drug development: fast, clean, and soft. Anesth Analg. 2012 Aug;115(2):220-2. doi: 10.1213/ANE.0b013e31825ef8d7. No abstract available. PMID 22826519
- [Background] Sear JW. Challenges of bringing a new sedative to market! Curr Opin Anaesthesiol. 2018 Aug;31(4):423-430. doi: 10.1097/ACO.0000000000000614. PMID 29847365
- [Background] Upton R, Martinez A, Grant C. A dose escalation study in sheep of the effects of the benzodiazepine CNS 7056 on sedation, the EEG and the respiratory and cardiovascular systems. Br J Pharmacol. 2008 Sep;155(1):52-61. doi: 10.1038/bjp.2008.228. Epub 2008 Jun 16. PMID 18552878
- [Background] Upton RN, Martinez AM, Grant C. Comparison of the sedative properties of CNS 7056, midazolam, and propofol in sheep. Br J Anaesth. 2009 Dec;103(6):848-57. doi: 10.1093/bja/aep269. Epub 2009 Sep 29. PMID 19797247
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Inouye SK, Schlesinger MJ, Lydon TJ. Delirium: a symptom of how hospital care is failing older persons and a window to improve quality of hospital care. Am J Med. 1999 May;106(5):565-73. doi: 10.1016/s0002-9343(99)00070-4. PMID 10335730
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Zaal IJ, Devlin JW, Hazelbag M, Klein Klouwenberg PM, van der Kooi AW, Ong DS, Cremer OL, Groenwold RH, Slooter AJ. Benzodiazepine-associated delirium in critically ill adults. Intensive Care Med. 2015 Dec;41(12):2130-7. doi: 10.1007/s00134-015-4063-z. Epub 2015 Sep 24. PMID 26404392
- [Background] Kassie GM, Nguyen TA, Kalisch Ellett LM, Pratt NL, Roughead EE. Preoperative medication use and postoperative delirium: a systematic review. BMC Geriatr. 2017 Dec 29;17(1):298. doi: 10.1186/s12877-017-0695-x. PMID 29284416
- [Background] Bohlken J, Kostev K. Prevalence and risk factors for delirium diagnosis in patients followed in general practices in Germany. Int Psychogeriatr. 2018 Apr;30(4):511-518. doi: 10.1017/S1041610217002587. Epub 2017 Dec 13. PMID 29235430
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Background] Yap A, Lopez-Olivo MA, Dubowitz J, Hiller J, Riedel B; Global Onco-Anesthesia Research Collaboration Group. Anesthetic technique and cancer outcomes: a meta-analysis of total intravenous versus volatile anesthesia. Can J Anaesth. 2019 May;66(5):546-561. doi: 10.1007/s12630-019-01330-x. Epub 2019 Mar 4. PMID 30834506